CLINICAL TRIAL: NCT02744274
Title: Randomized, Assessor- and Participant-blinded, Controlled, and Parallel-design Approach to Investigate Whether Acupuncture Can Prevent or Postpone the Occurrence of Peripheral Neuropathy and Improve Quality of Life.
Brief Title: Efficacy of Acupuncture in Prevention of Chemotherapy Induced Peripheral Neuropathy - a Pilot Study
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tzu-Liang Chen (Other)
Collaborators: Research Center For Chinese Medicine and Acupuncture (Unknown)
Responsible Party: Sponsor-Investigator, Tzu-Liang Chen, Deputy Superintendent of the Surgery department, China Medical University Hospital
Organization: China Medical University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CMUH104-REC1-076
Record Dates: First submitted 2016-04-13; First posted 2016-04-20 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Colorectal Cancer
Keywords: acupuncture; chemotherapy; peripheral neuropathy; randomized clinical trial; numbness
MeSH Terms: conditions — Colorectal Neoplasms; Peripheral Nervous System Diseases; Hypesthesia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Verum acupuncture (Experimental): 16 patients will be randomized to receive verum acupuncture two times biweekly, prior to beginning chemotherapy and the weeks that drugs administered, for 26 treatments in total.
  Interventions: Other: Verum acupuncture
- Sham acupuncture (Placebo Comparator): 16 patients will be randomized to receive sham acupuncture two times biweekly, prior to beginning chemotherapy and the weeks that drugs administered, for 26 treatments in total.
  Interventions: Other: Verum acupuncture

INTERVENTIONS:
Other: Verum acupuncture — Patients will lay supine. The acupuncture physicians will disinfect the selected acupuncture points with alcohol and then needle them (30 gauze, 1.5-inch, Yuguang, Taiwan) with a plastic device is fixed needle body, so that the patient achieves a "de qi" sensation, which is often described as a pressure or achiness feeling. The acupuncture point will be bilateral Quchi, Waiguan, hegu, baxie, Zusanli, Yanglingquan, Sanyinjiao, Taichong, bafeng. Acupuncture needles will be left in place for approximately 30 minutes, and every 10 minutes twisting stainless steel needle to get a "de qi".

SUMMARY:
The aim of this pilot study is to investigate the efficacy of acupuncture in prevention of chemotherapy induced peripheral neuropathy. The study adapted a single center, randomized, assessor- and participant-blinded, controlled, and parallel-design approach to investigate whether acupuncture can prevent or postpone the occurrence of peripheral neuropathy and improve quality of life.

DETAILED DESCRIPTION:
Background and purpose:

Chemotherapy-induced peripheral neuropathy (CIPN) is a disabling side effect of several commonly used antineoplastic agents. CIPN prevalence was 68.1% within the first month of the end of chemotherapy, 60% at 3 months, and 30.0% at 6 months or later. Oxaliplatin as a chemotherapeutic drug for colorectal cancer has neurotoxicity on peripheral nerve system. A definite portion of patients suffered neurologic symptoms including paresthesia, dysesthesia over limbs and perioral area accompanied with muscles cramps or spasm sometimes; however, had impact on quality of life, daily functions, quality of sleep and lead to distress and depression. There is no drug to prevent peripheral neuropathy. Clinical observations reveal that acupuncture could decrease peripheral neuropathy, improve quality of life, and promote motivation of complete chemotherapy course.

Material and methods:

A total of 32 volunteers of patients with colorectal cancer will be recruited from the Chinese medicine or Western medicine clinics in China Medical University Hospital. These patients will be randomized to receive verum acupuncture or sham acupuncture treatment two times biweekly, prior to beginning chemotherapy and the weeks that drugs administered, for 26 treatments in total.

Questionnaires, neurological examination and Von Frey Filament Test will be completed at baseline, 12 and 24 weeks after initiation of intervention, 12 and 24 weeks after completion of acupuncture completion.

Predict results:

Investigators expect that the efficacy of verum acupuncture is superior to sham acupuncture in prevent or postpone occurrence of chemotherapy induced peripheral neuropathy and able to improve numbness, paresthesia, quality of life. The effectiveness of acupuncture can be detected by questionnaires, Von Frey Filament Test and neurological testing.

ELIGIBILITY:
Inclusion Criteria:

1. Patients were diagnosed as stage 3 colorectal cancer.
2. Patients are going to receive Oxaliplatin based chemotherapy.
3. Patients are willing to cooperate with physicians and completely receive chemotherapy.
4. Patients are willing to receive acupuncture treatments and follow-up assessments.
5. Adult volunteers with the ages of 20-70 years old.
6. ECOG Performance Status of 0, 1, or 2

Exclusion Criteria:

1. Current active treatments with chemotherapy, radiotherapy or tumor resection surgery in the past one month.
2. Having chemotherapy with neuropathic agents including taxane, platinum, vinca alkaloid, bortezimab, or thalidomide in the past six months.
3. Local infection at or near the acupuncture site is not suitable for acupuncture after physician examination.
4. Concurrent use of other alternative medicines such as herbal agents, high dose vitamins and minerals.
5. Known coagulopathy or taking anticoagulants.
6. Platelets < 50000/ul.
7. WBCs < 3000/ul.
8. Active CNS disease
9. Cardiac pacemaker.
10. Psychological or behavior disorder such as Schizophrenia.
11. Currently pregnant or breastfeeding women.
12. History of diabetic neuropathy or neuropathy related to HIV.
13. Previous acupuncture treatment for any indication within 30 days of enrollment.
14. Current medications that could affect symptoms related to CIPN.
15. Grade III lymphedema or more severe situation

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in NCV at 48weeks. | Baseline, 12 and 24 weeks after initiation of intervention, 12 and 24 weeks after completion of acupuncture completion.
Change from Baseline in Von frey filament test at 48weeks. | Baseline, 12 and 24 weeks after initiation of intervention, 12 and 24 weeks after completion of acupuncture completion.

SECONDARY OUTCOMES:
Change from Baseline in questionnaire - FACT/GOG-Ntx Subscale at 48weeks. | Baseline, 12 and 24 weeks after initiation of intervention, 12 and 24 weeks after completion of acupuncture completion.
Change from Baseline in questionnaire - FACT-G at 48weeks. | Baseline, 12 and 24 weeks after initiation of intervention, 12 and 24 weeks after completion of acupuncture completion.
Change from Baseline in questionnaire - Brief Pain Inventory Short Form at 48weeks. | Baseline, 12 and 24 weeks after initiation of intervention, 12 and 24 weeks after completion of acupuncture completion.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided